CLINICAL TRIAL: NCT05749562
Title: Study of the Effect of a Cheneau-Toulouse-Munster Brace in the Treatment of Adolescent Idiopathic Scoliosis on Respiratory Function
Brief Title: Effect of a Brace on the Adolescent Idiopathic Scoliosis Breathing
Acronym: CTM biomec
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO23019*
Record Dates: First submitted 2023-02-06; First posted 2023-03-01 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Adolescent; Female; Biomechanical Phenomena

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescent Idiopathic Scoliosis with right thoracic or thoraco-lumbar curvature: Patients will be treated with a Cheneau-Toulouse-Munster (CTM) brace, with a wearing time of more than 12 hours/24h, for more than 1 month.
  Interventions: Device: Cheneau-Toulouse-Munster brace

INTERVENTIONS:
Device: Cheneau-Toulouse-Munster brace — Full length, orthogonal anteroposterior and lateral X-rays will be taken with the Cheneau-Toulouse-Munster brace.

SUMMARY:
This study intends to investigate the effect of bracing on respiratory function in the treatment of adolescent idiopathic scoliosis (AIS). In particular, it will look at the effect of the brace on respiratory function and 3D volume of the thoracic cage. An additional evaluation of the pressure forces of the brace, using a connected t-shirt, will be carried out. The investigators hypothesise that the brace will decrease the respiratory parameters and 3D volume of the thoracic cage, especially during deep breathing.

DETAILED DESCRIPTION:
Scoliosis is a 3D deformity of the spine with curvatures occurring in the three planes of space.

The brace is widely used for adolescent idiopathic scoliosis. The Cheneau-Toulouse-Munster (CTM) brace is a rigid brace, classically indicated for thoracic and lumbar curves. However, scoliosis induces structural deformation of the rib cage. This can lead to changes in thoracic volume associated with a respiratory disorder, mainly restrictive. But the effect of bracing on pulmonary function currently remains unclear.

Few studies in the literature have looked at the impact of the brace on lung function. In those studies, the findings were based on Pulmonary Function Test (PFT) results only. In the CTM biomec study, the investigators propose to evaluate lung function by PFT associated with biplanar radiography using EOS® system, which allows 3D modelling of the rib cage. An additional evaluation of the pressure forces of the CTM brace, using a connected t-shirt, will be carried out to better understand the biomechanics of the brace. It will allow us to observe the stress surfaces on the thorax during the respiratory cycle and to compare them with the adaptation kinematics of the thoracic cage.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent girls aged 12 to 16
* With a right thoracic or thoraco-lumbar curvature (right and left)
* With a Cobb angle between 20 and 40°.
* Treated with a Cheneau-Toulouse-Munster brace for more than 1 month
* With a duration of brace wearing of more than 12/24h
* Affiliated to a social security system

Exclusion Criteria:

* Male gender
* Having a secondary scoliosis (neuromuscular, syndromic, post-traumatic, congenital pathology)
* Having a respiratory pathology prior to the diagnosis of scoliosis
* Have a history of spinal surgery
* Having already benefited from a brace treatment

Ages: 12 Years to 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Study Population: The study will be conducted with patients treated for scoliosis in the Department of Pediatric Surgery, at the American Memorial Hospital, CHU Reims.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2023-02-17 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
Total Lung Capacity (TLC) | 1 day
  change with and without the brace

SECONDARY OUTCOMES:
Forced expiratory volume in one second | 1 day
  change with and without the brace

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided